CLINICAL TRIAL: NCT05789680
Title: European Multicentric Study on Parathyroid Carcinoma
Acronym: EMS-PC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 5287
Record Dates: First submitted 2023-03-16; First posted 2023-03-29 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-02

CONDITIONS: Parathyroid Carcinoma
Keywords: parathyroid carcinoma; primary hyperparathyroidism; Eurocrine
MeSH Terms: conditions — Parathyroid Neoplasms; Hyperparathyroidism, Primary | interventions — Parathyroidectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Parathyroid carcinoma among patients undergoing surgical treatment of primary hyperparathyroidism: All adult (18 years old and older) patients registered in EUROCRINE® database that underwent surgery for primary hyperparathyroidism and received histopathologic diagnosis of parathyroid carcinoma from 2015 till 2021 will be included
  Interventions: Procedure: Surgical treatment of parathyroid carcinoma

INTERVENTIONS:
Procedure: Surgical treatment of parathyroid carcinoma — Radical treatment of suspected parathyroid carcinoma should consist of parathyroidectomy and en bloc ipsilateral hemithyroidectomy and central lymph node dissection.
  Other Names: parathyroidectomy; ipsilateral hemithyroidectomy; ipsilateral central neck dissection

SUMMARY:
The main aim of the study is to evaluate the incidence of post-operative diagnosis of PC and atypical parathyroid neoplasm in patients who underwent surgery for pHPT in different European centers using the EUROCRINE® database. Moreover, we aim to evaluate the peri-operative surgical characteristics, operation extent, postoperative morbidity, and outcomes in these patients category.

DETAILED DESCRIPTION:
Parathyroid cancer (PC) is one of the rarest malignancies (0.005% of all tumours) and it represents less than 1% of all the causes of primary hyperparathyroidism (pHPT).

It is frequently a sporadic disease, but it can be part of hereditary syndromes (i.e. HPT- JT, MEN, MEN2A and FIHP).

Clinical and biochemical presentation is usually more severe comparing to other forms of primary hyperparathyroidism as it is often associated to very high serum-calcium and PTH levels and target organs' damages.

Malignancy should be suspected on the basis of the aforementioned biochemical data and the imaging evidences (such as parathyroid lesion dimension >3 cm, faded edges, inhomogeneous internal features and cervical lymph nodes enlargement).

In case of suspected PC a radical treatment should be proposed to the patient, consisting of parathyroidectomy and en bloc ipsilateral hemithyroidectomy and ipsilateral central neck dissection. Indeed, the oncological radicality during surgical treatment is mandatory, as effective adjuvant therapy is not available.

However, pre-operative differential diagnosis with parathyroid adenoma is still challenging, thus malignancy can be detected only after the histological analysis of the specimen and sometimes after recurrences.

Moreover, parathyroid atypical adenoma entity is still controversial, as it presents suspicious histological features, but certain signs of malignancy are lacking (such as capsular, vessels and neural invasion). Furthermore, natural history and biological behaviour are still unknown.

ELIGIBILITY:
Inclusion Criteria: All adult (18 years old and older) patients that underwent surgery for primary hyperparathyroidism with a final histology of parathyroid carcinoma from 2015 till 2021.

Inclusion Criteria:

* All adult (18 years old and older) patients
* underwent surgery
* final histology of parathyroid carcinoma
* among European centers that participate in the Eurocrine® database between 2015 and 2021

Exclusion Criteria:

• Patients <18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with final histology of parathyroid carcinoma operated among European centers that participate in the Eurocrine® database between 2015 and 2021
Sampling Method: Non-Probability Sample
Enrollment: 17 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of parathyroid carcinoma | January 2015-January 2021
  Descriptive analysis of the exact incidence of parathyroid carcinoma among patients undergoing surgical treatment of primary hyperparathyroidism in European centers.

SECONDARY OUTCOMES:
Oncologic outcome | January 2015-January 2021
  Descriptive analysis of operative and oncologic outcome of patients undergoing surgical treatment of primary hyperparathyroidism and receiving pathological report od parathyroid carcinoma in European centers.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Raffaelli, Prof, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Reasonable requests will be evaluated by the Eurocrine Council